CLINICAL TRIAL: NCT00013897
Title: A Phase III Study Comparing the Antiviral Efficacy and Safety of BMS-232632 With Efavirenz; Each in Combination With Fixed Dose Zidovudine-Lamivudine
Brief Title: A Comparison of BMS-232632 With Efavirenz, Each in Combination With Zidovudine-Lamivudine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 302C; AI424-034
Record Dates: First submitted 2001-03-31; First posted 2001-08-31 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: Placebos; Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; BMS 232632; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; lamivudine, zidovudine drug combination; efavirenz

INTERVENTIONS:
Drug: Atazanavir
Drug: Lamivudine/Zidovudine
Drug: Efavirenz

SUMMARY:
The purpose of this study is to compare the effectiveness of treatment with BMS-232632 to that of efavirenz (EFV) when both are used with zidovudine (ZDV) and lamivudine (3TC).

DETAILED DESCRIPTION:
This is a multinational, 2-arm study. Patients in 1 arm receive BMS-232632 plus EFV placebo capsules. Patients in the other arm receive EFV plus BMS-232632 placebo. Both arms also receive a fixed dose of ZDV-3TC.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have a viral load of 2,000 or more copies/ml and a CD4 cell count of 100 or more cells/mm3 (or 75 or more cells/mm3 with no prior history of AIDS-defining diagnosis) within 2 weeks before randomization.
* Are at least 16 years old.
* Have signed consent of parent or guardian if under 18 years of age.
* Are willing to use effective barrier methods of birth control.
* Are available for follow-up for at least 52 weeks.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have had anti-HIV treatment within 30 days before screening.
* Have a recently diagnosed HIV-related infection.
* Have any medical condition requiring treatment at enrollment.
* Have recently become HIV infected.
* Have acute hepatitis within 30 days of study entry. Certain patients with chronic hepatitis will be eligible.
* Expect to need or have taken drugs with myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic, or cytotoxic potential within 3 months before study. Expect to need methadone, ribavirin/interferons, neurotoxic drugs or drugs that affect CYP3A4.
* Abuse alcohol or drugs.
* Have severe diarrhea within 30 days before study entry.
* Are pregnant or breast-feeding.
* Have a history of hemophilia.
* Have a history of bilateral peripheral neuropathy.
* Cannot take medicines by mouth.
* Have any other conditions that the doctor thinks would interfere with the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (99):
- United States (28):
  - Phoenix Body Positive, Phoenix, Arizona
  - Univ of Southern California, Los Angeles, California
  - Saint Francis Mem Hosp / HIV Care Unit, San Francisco, California
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Dr Bruce Rashbaum, Washington D.C., District of Columbia
  - North Broward Hosp District / HIV Clinical Research, Fort Lauderdale, Florida
  - Associates in Research, Fort Myers, Florida
  - Steinhart Medical Associates, Miami, Florida
  - Saint Josephs Comprehensive Research Institute, Tampa, Florida
  - Emory Univ, Atlanta, Georgia
  - The CORE Ctr, Chicago, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Univ of Michigan Hospitals and Health Ctrs, Ann Arbor, Michigan
  - Washington Univ School of Medicine, St Louis, Missouri
  - Univ of Nebraska Medical Ctr, Omaha, Nebraska
  - Robert Wood Johnson Med School/UMDNJ, New Brunswick, New Jersey
  - UMDNJ - New Jersey Med School, Newark, New Jersey
  - ID Care Inc, Somerville, New Jersey
  - Univ of NM, Albuquerque, New Mexico
  - Duke Univ Med Ctr / Infectious Disease Clinic, Durham, North Carolina
  - Jemsek Clinic, Huntersville, North Carolina
  - Ohio State Univ Hosp, Columbus, Ohio
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Methodist Healthcare, Memphis, Tennessee
  - Oaklawn Physicians Group, Dallas, Texas
  - Tarrant County Infectious Diseases Associates, Fort Worth, Texas
  - Montrose Clinic, Houston, Texas
- Austria (2):
  - AKH Wien, Vienna
  - Pulmologisches Zentrum Der Stadt Wien, Vienna
- Belgium (2):
  - CHU Saint Pierre, Brussels
  - UZ Gasthuisberg, Leuven
- Canada (4):
  - Univ of Alberta/Division of Inf Dis/Dept of Med, Edmonton, Alberta
  - Univ of British Columbia, Vancouver, British Columbia
  - McMaster Univ Med Ctr, Hamilton, Ontario
  - Gary Rubin, Toronto, Ontario
- Chile (4):
  - Fundacion Arriaran, Santiago
  - Hosp Clinico de La Pontificia Universidad Catolica de Chile, Santiago
  - Hosp Sotero de Rio, Santiago
  - Servicio de Dermatologia-Hosp del Salvador, Santiago
- SEMECO, San José, Costa Rica
- France (5):
  - Hopital Hotel Dieu de Lyon, Lyon
  - CHU De Bicetre, Paris
  - Hopital Cochin - Port Royal, Paris
  - Services des Maladies Infectieuses, Paris
  - Hospital Gustave Dron, Tourcoing
- Germany (2):
  - Rheinische Friedrich Wilhelms Universitaet Medizinische, Bonn
  - Univ Zu Koeln, Cologne
- Guatemala (2):
  - Hosp General San Juan de Dios, Guatemala City
  - Hosp Roosevelt Chief Infectious Diseases Unit, Guatemala City
- Saint Laszlo Hosp, Budapest, Hungary
- Kaplan Med Ctr, Rehovot, Israel
- Italy (8):
  - Ospedale S Orsola, Bologna
  - Immunoligia Universita Cagliari, Cagliari
  - Ospedale Luigi Sacco Cargnel, Milan
  - Ospedale S Raffaele, Milan
  - Ospedale degli Infermi, Rimini
  - Cat All Immun Clin, Roma
  - Ospedale Amedeo de Savoia, Torino
  - Ospedale Amedeo di Savoia, Torino
- Malaysia (2):
  - Hosp Kuala Lumpur, Kuala Lumpur
  - Univ of Malaya Med Ctr, Kuala Lumpur
- Consultorio Royal Ctr, Panama City, Panama
- Peru (5):
  - Hosp Edgardo Rebagliati, Lima
  - Hosp Guillermo Almenara-Medicina 1, Lima
  - Hosp Nacional Arzobispo Loayza-PROCETS, Lima
  - Hosp Nacional Cayetano Heredia, Lima
  - Hosp Nacional dos de Mayo, Lima
- Portugal (2):
  - Hosp De Santa Maria, Lisbon
  - Hosp De Sao Joao, Porto
- Puerto Rico (2):
  - Clinical Research Puerto Rico Inc, San Juan
  - San Juan VAMC, San Juan
- Russia (3):
  - Federal AIDS Ctr, Moscow
  - Infectious Hosp 30, Saint Petersburg
  - Ust Izhora Fed Infectious Hosp, Saint Petersburg
- South Africa (4):
  - Brooklyn Med Ctr, Cape Town
  - Tygerberg Hosp, Cape Town
  - Chris Hani Baragwanath Hosp, Johannesburg
  - Toga Lab, Johannesburg
- Spain (8):
  - Hosp Clinic, Barcelona
  - Hosp Germans Trias I Pujol, Barcelona
  - Hosp de Basurto / Enfermedades Infecciosas, Bilboa
  - Hosp Reina Sofia, Córdoba
  - Hosp Carlos III, Madrid
  - Hosp Ramon y Cajal, Madris
  - Hosp Nuestra Senora de Covadonga, Oviedo
  - Hosp Virgen Del Rocio, Seville
- Universitatsspital Zurich, Zurich, Switzerland
- Thailand (5):
  - Rajavithi Hosp, Bangkok
  - Ramathibodi Hosp, Bangkok
  - Siriraj Hosp / Mahidol Univ, Bangkok
  - Vajira Hosp, Bangkok
  - Chiangmai Univ, Chiang Mai
- United Kingdom (3):
  - King's College Hosp, Cambewell
  - Saint James Hosp, Dublin
  - Royal Free Hosp, London
- Venezuela (3):
  - Hosp U de Caracas / Ciudad, Caracas
  - Hosp Vargas de Caracas, Caracas
  - Hosp Dr Domingo Luciani, Miranda